CLINICAL TRIAL: NCT00643227
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Comparative Trial of Azithromycin SR Versus Clarithromycin Extended Release for the Treatment of Mild to Moderate Community-Acquired Pneumonia in Adults
Brief Title: A Multicenter, Randomized, Double-Blind, Double-Dummy Trial of Azithromycin SR Compared With Clarithromycin Extended Release for the Treatment of Pneumonia in Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Diretor, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661075
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2008-03-26 (Estimated); Status verified 2008-03

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: clarithromycin extended release (ER)
- 2 (Experimental)
  Interventions: Drug: azithromycin SR

INTERVENTIONS:
Drug: clarithromycin extended release (ER) — 7 days of clarithromycin extended release (ER), 1.0 g by mouth once daily
  Arms: 1
Drug: azithromycin SR — Single, 2.0 g oral dose of azithromycin sustained release (SR) by mouth once daily
  Arms: 2

SUMMARY:
The study was performed to confirm that a single, 2.0 g oral dose of azithromycin sustained release (SR) at least as effective as 7 days of clarithromycin extended release (ER), 1.0 g by mouth once daily, when used to treat adults with mild to moderate community acquired pneumonia (CAP), and that both treatments were safe.

ELIGIBILITY:
Inclusion Criteria:

Outpatients with a diagnosis of pneumonia, as demonstrated by a productive cough and at least 2 of the following signs and symptoms: rales and/or evidence of pulmonary consolidation; dyspnea or tachypnea; elevated body temperature; or elevated total peripheral white blood cell count (WBC >10,000/mm3) or greater than 15% immature neutrophils were included. Patients were to have a chest radiograph demonstrating evidence of a new infiltrate or consolidation, and a Modified Fine Risk score of ≤ 70 (Fine Class I and II).

Exclusion Criteria:

Patients who were treated with any systemic antibiotic of greater than 1 dose or 1 combination dose (such as cephalosporin and macrolide) within the previous 7 days, or the likelihood of receiving other systemic antibiotics during participation in the study; were hospitalized in the previous 14 days or had an infection acquired in the hospital, and who were residents of a long-term care facility were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2003-01; Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
sponsor assessment of clinical response (clinical cure rate) in the Clinical Per Protocol population | Test of Cure (TOC) visit (Day 14-21)

SECONDARY OUTCOMES:
bacteriologic response (eradication rate) in the Bacteriological Per Protocol population | TOC visit
investigator assessment of clinical response in the Clinical Per Protocol population | TOC visit
sponsor assessment of clinical response by baseline pathogen | End of Treatment (EOT) visit (Day 8-11) and TOC visit
sponsor assessment of clinical response in the non-primary population | EOT visit and TOC visit
sponsor assessment of clinical responses in the Clinical Per Protocol population | EOT visit and Long-Term Follow-Up (LTFU) visit (Day 28-35)
susceptibilities of baseline pathogens | Study endpoint
adverse events | Continuous
vital signs | Baseline, On-Treatment (OT) visit (Day 3-5), and TOC visit
physical examination | Baseline
clinical laboratory assessments (blood chemistry and hematology) | Baseline and TOC visit

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- United States (27):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Haleyville, Alabama
  - Pfizer Investigational Site, Montgomery, Alabama
  - Pfizer Investigational Site, Tallassee, Alabama
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tempe, Arizona
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Boise, Idaho
  - Pfizer Investigational Site, Meridian, Idaho
  - Pfizer Investigational Site, Nampa, Idaho
  - Pfizer Investigational Site, Chalmette, Louisiana
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Butte, Montana
  - Pfizer Investigational Site, Holmdel, New Jersey
  - Pfizer Investigational Site, Clemmons, North Carolina
  - Pfizer Investigational Site, Salisbury, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Summerville, South Carolina
  - Pfizer Investigational Site, Milan, Tennessee
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Taylorsville, Utah
  - Pfizer Investigational Site, West Jordan, Utah
  - Pfizer Investigational Site, Casper, Wyoming
- Argentina (2):
  - Pfizer Investigational Site, Tandil, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires
- Canada (12):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, St. John's, Newfoundland and Labrador
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Drummondville, Quebec
  - Pfizer Investigational Site, Granby, Quebec
  - Pfizer Investigational Site, Longueuil, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Saint-Jérôme, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec
  - Pfizer Investigational Site, Saskatoon, Saskatchewan
- Estonia (2):
  - Pfizer Investigational Site, Tallinn
  - Pfizer Investigational Site, Tartu
- India (6):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Elamakkara, Cochin, Kerala
  - Pfizer Investigational Site, Pune, Maharashtra
  - Pfizer Investigational Site, Ludhiana, Punjab
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
- Lithuania (2):
  - Pfizer Investigational Site, Kaunas
  - Pfizer Investigational Site, Vilnius
- Russia (2):
  - Pfizer Investigational Site, Moscow
  - Pfizer Investigational Site, Smolensk
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661075&StudyName=A%20Multicenter%2C%20Randomized%2C%20Double-Blind%2C%20Double-Dummy%20Trial%20of%20Azithromycin%20SR%20Compared%20with%20Clarithromycin%20Extended%20Release%20for%20the%20Tre